CLINICAL TRIAL: NCT01911897
Title: CALM-FIM_EUR - Controlling and Lowering Blood Pressure With the MobiusHD - A Prospective Multicenter Safety Study
Brief Title: Controlling and Lowering Blood Pressure With The MOBIUS HD™ (CALM-FIM_EUR)
Acronym: CALM-FIM_EUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD0120, CRD0233
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MobiusHD (Experimental): MobiusHD
  Interventions: Device: MobiusHD

INTERVENTIONS:
Device: MobiusHD — Implant that is placed in the carotid sinus to control hypertension.

SUMMARY:
To evaluate the safety and performance of the MobiusHD system in subjects with resistant hypertension.

DETAILED DESCRIPTION:
This is an open-label, multicenter, first-in-man clinical trial to be conducted in Europe. Eligible subjects with stage 2 resistant systemic arterial hypertension currently being treated with a minimum of three (3) anti-hypertensive drugs, who consent to study participation will be assigned to treatment with the MobiusHD system.

Potential study participants will be consented and then screened at two (2) baseline visits beginning at least 30 days prior to MobiusHD placement. Qualified patients will undergo placement of the MobiusHD under angiographic visualization, and will then be followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Office cuff SBP ≥ 160 mmHg measured per protocol instructions following at least one (1) month of maximally tolerated therapy with at least three (3) anti-hypertensive medications, of which at least one (1) must be a diuretic unless patient has history of intolerance, ineffectiveness or contraindications.

Exclusion Criteria:

* Known or clinically suspected baroreflex failure or autonomic neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van der Heyden, MD, Principal Investigator — St. Antonius Hospital
Locations (6):
- University of Cologne, Cologne, Germany
- Netherlands (5):
  - Maastricht University Medical Center, Maastricht, AZ
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Kleef MEAM, Devireddy CM, van der Heyden J, Bates MC, Bakris GL, Stone GW, Williams B, Spiering W; CALM-FIM Investigators. Treatment of Resistant Hypertension With Endovascular Baroreflex Amplification: 3-Year Results From the CALM-FIM Study. JACC Cardiovasc Interv. 2022 Feb 14;15(3):321-332. doi: 10.1016/j.jcin.2021.12.015. PMID 35144789
- [Derived] Spiering W, Williams B, Van der Heyden J, van Kleef M, Lo R, Versmissen J, Moelker A, Kroon A, Reuter H, Ansel G, Stone GW, Bates M; CALM-FIM_EUR investigators. Endovascular baroreflex amplification for resistant hypertension: a safety and proof-of-principle clinical study. Lancet. 2017 Dec 16;390(10113):2655-2661. doi: 10.1016/S0140-6736(17)32337-1. Epub 2017 Sep 1. PMID 28870716
- [Derived] Habib N, Mahmoodi BK, Bos WJ, Tromp SC, Suttorp MJ, Bates MC, Van der Heyden J. Initial experience with therapeutic geometric modification of the carotid bulb for true resistant hypertension. EuroIntervention. 2015 May;11(1):117-20. doi: 10.4244/EIJV11I1A20. PMID 25982654

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MobiusHD
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | MobiusHD
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  Germany | 28
Systolic Office Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 184 (18.4)
24-Hour Ambulatory Blood Pressure (Systolic Blood Pressure) [Mean (Standard Deviation); unit: mmHg] — Ambulatory blood pressure monitoring (ABPM) is a method to measure blood pressure on a continuous basis for 24 hours. Ambulatory blood pressure monitoring is accomplished with a special device that consists of a blood pressure cuff worn on the arm. It's attached to a small recording device that the patient wears. The ABPM device is worn for 24 hours.
  mmHg | 167 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The number of participants with serious adverse events reported in the study will be tabulated.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | MobiusHD
Number analyzed (Participants) | 30
Participants | 8

2. Secondary Outcome: Systolic Office Cuff Blood Pressure (BP)
Time Frame: Baseline, discharge (up to 2 days), 7 days, 1 month, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MobiusHD
Number analyzed (Participants) | 30
mmHg
  Baseline | 184 (18.4)
  Discharge (up to 2 days) | 147 (22.2)
  7 days | 157 (27.3)
  1 month | 162 (30.6)
  3 months | 160 (28.4)
  6 months | 160 (26.1)

3. Secondary Outcome: Mean 24-hour Systolic Ambulatory Blood Pressure (ABPM) at 6 Months
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MobiusHD
Number analyzed (Participants) | 30
mmHg
  Baseline | 167 (16.6)
  3 months | 150 (19.1)
  6 months | 145 (19.1)

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | MobiusHD
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MobiusHD (N=30)
Hypertensive Emergency (Cardiac disorders) | 2 (2)
Hypotension - chronic (Cardiac disorders) | 2 (2) — Chronic = more than 30 days post procedure
Relative hypotension - acute (Cardiac disorders) | 1 (1) — Acute = 1-7 days post procedure
Stroke with permanent symptoms (General disorders) | 1 (1)
Transient ischemic attack (General disorders) | 1 (1)
Access site complications (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MobiusHD (N=30)
Access site complications (General disorders) | 5 (5)
Dizziness (General disorders) | 6 (6)
Hypotension - acute (Cardiac disorders) | 2 (2) — Acute = 1-7 days post procedure
Pain (General disorders) | 8 (9)
Relative hypotension - acute (Cardiac disorders) | 2 (2) — Acute = 1-7 days post procedure
Skin sensation disturbance (General disorders) | 3 (3)
Transient ischemic attack (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No